CLINICAL TRIAL: NCT01120262
Title: Germline Polymorphisms Associated With the PSA Response in Men With Metastatic Prostate Cancer Treated With Androgen Deprivation Therapy
Brief Title: S9346A Blood Samples From Patients With Metastatic Prostate Cancer Previously Treated With Bicalutamide and Goserelin
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000669307; SWOG-S9346A
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is studying blood samples from patients with metastatic prostate cancer previously treated with bicalutamide and goserelin.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the association between serum PSA response (< 4 ng/mL) at 7 months with inherited variability of germline single nucleotide polymorphisms, in a set of candidate genes, in patients with metastatic prostate cancer treated with combination induction androgen-deprivation therapy comprising bicalutamide and goserelin.

OUTLINE: DNA extracted from whole blood or serum samples is analyzed for inherited variability of germline single nucleotide polymorphisms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with metastatic prostate cancer
* Accrued to SWOG-9346 and received androgen-deprivation therapy (ADT)
* Must have serum PSA values from the beginning to the end of 8 courses of ADT
* Must have whole blood or serum samples available

PATIENT CHARACTERISTICS:

* Caucasian and African-American participants

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: S9346 patients
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Serum PSA values at 7 months | 7 months
Role of genetic variation in response to therapy | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A. Cooney, MD, Principal Investigator — University of Michigan Rogel Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf